CLINICAL TRIAL: NCT04806815
Title: Menstrual Cycle-induced Pain, Fatigue and Anxiety in Women Suffered From COVID-19
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Associated Proffesor, Biruni University
Other Study IDs: 2021/47-45
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Menstrual Problem; Covid19; Fatigue
Keywords: Menstrual Problem; Covid19; Fatigue
MeSH Terms: conditions — Menstruation Disturbances; COVID-19; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A survey of 60 questions was created through the internet-based 'Google Forms surveys' site. — The following tests will be used together with the survey;
  * Menstrual Symptom Questionnaire
  * Fatigue Severity Scale
  * Short Form Of Coronavirus Anxiety Scale

SUMMARY:
The effects of COVID-19 on body systems and functions are still being investigated. ACE 2, which plays a key role in the entry of the COVID-19 virus into the cell, is also highly expressed in the ovary, uterus, vagina, and placenta in the female genital system, which can also pose a risk to female reproductive health. The aim of this study is to evaluate menstrual cycle-induced pain, fatigue and anxiety in women who suffered from COVID-19.

DETAILED DESCRIPTION:
The effects of COVID-19 on body systems and functions are still being investigated. ACE 2, which plays a key role in the entry of the COVID-19 virus into the cell, is also highly expressed in the ovary, uterus, vagina, and placenta in the female genital system, which can also pose a risk to female reproductive health. It has been examined that menstruation volume decreased or cycle lengthened in one-fifth of women who had COVID-19, and this condition was more intense in those who had severe COVID-19. Studies have shown that the possible effects of COVID-19 on the female genital system often remain theoretical hypotheses. In the literature, there was no study in which menstrual dysfunctions and secondary problems caused by the state of inactivity entering our lives during pandemic were discussed in a wide spectrum of women who had COVID-19. Therefore the aim of this study is to evaluate menstrual cycle-induced pain, fatigue and anxiety in women who suffered from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 45,
* PCR test result positive confirmed having COVID-19 infection,
* Women had at least one period of Menstrual cycle after COVID-19
* Being an Internet connection,
* To be able to speak and write in Turkish.

Exclusion Criteria:

* To be in the premenaposual/postmenopausal period (to be in the transition period to menopause or in the period after menopause.)
* Having insufficient co-operation.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female individuals aged 18-45 who have had COVID-19
Study Population: The study will include 200 volunteers, female individuals aged 18-45 who have had COVID-19.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Menstrual Symptom Questionnaire | 1 day
  This scale was developed to assess menstrual pain and symptoms. It is a five-point Likert-type scale consisting of 24 items. Participants will be asked to give a number between 1 (never) and 5 (always) to their menstrual symptoms. Total score will be calculated by taking the total score of the items in the scale. Increasing the average score indicates that the severity of menstrual symptoms increased.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 1 day
  Each question in this scale consisting of Likert type questions: (1) I strongly disagree (2) I do not attend (3) I tend not to participate (4) I am indecisive (5) I tend to join (6) I participate (7) It is scored as I strongly agree. A score of 4 or higher on the questions indicates severe fatigue. The scoring of the scale, which consists of 9 questions in total, varies between 9 and 63, while a total score of 36 and above indicates fatigue.
Short Form Of Coronavirus Anxiety Scale | 1 day
  The questionnaire has a five-point Likert type rating and consists of 5 items. "0: none", "1: rarely, less than a day or two", "2: a few days", "3: more than 7 days," They will be asked to rank the options "," 4: almost every day during the last two weeks "according to the five elements of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, Study Director — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)